CLINICAL TRIAL: NCT00385099
Title: A Phase IIa Pharmacodynamic Study of Antagonism of Irritable Bowel Syndrome (IBS) Symptoms by GW876008, a Corticotrophin Releasing Factor 1 Receptor Antagonist (CRF1-RA)
Brief Title: Effects Of GW876008 On The Bowel In Patients With Irritable Bowel Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Purpose: Treatment
Other Study IDs: CRI103143
Record Dates: First submitted 2006-10-04; First posted 2006-10-06 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Irritable Colon
Keywords: IBS; stress; CRF1
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — GW 876008

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GW876008

SUMMARY:
The purpose of this study is to see if GW876008 in Irritable Bowel Syndrome patients will reverse stress-induced hypersensitivity, by looking at thresholds for perception and pain.

ELIGIBILITY:
Inclusion criteria:

* Must have irritable bowel syndrome.

Exclusion criteria:

* Subjects who have been taking any medication for the treatment of irritable bowel syndrome within 6 months prior to the start of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-12-08 (Actual); Primary Completion 2007-10-15 (Actual); Study Completion 2007-10-15 (Actual)

PRIMARY OUTCOMES:
Percent change from Baseline in Laser Doppler regional Rectal Mucosal Blood Flow (RMBF) measured in response to physiological stress (cold water pressor test) | Baseline (pre-dose) and Study Days 1, 2 and 3
  Laser Doppler flowmetry measures changes in red cell flux using a probe that scans a fixed volume of tissue. Participants were examined in the left lateral position where DRT4 laser Doppler flow meter was placed against the rectal mucosa 10 centimeter (cm) above the lower limit of the anal margin, and pre-stress readings were taken after a period of 10 minutes of acclimatization in a room with an ambient temperature of 22 degrees Celsius. Physiological stress was evoked using the cold water pressor test. Participants were asked to place their hand and forearm into a container of ice-cold water at 0-4degree Celsius and were persuaded to maintain that position for as long as possible during the stress period of 10 minutes. Readings were then taken during pre-stress and at 5-minute intervals during the stress and recovery periods. Baseline was defined as the pre-dose assessment. Change from Baseline was calculated by subtracting the Baseline value minus the post-randomization value.
Percent Change from Baseline in Laser Doppler regional RMBF measured in response to psychological stress (dichotomous listening test) | Baseline (pre-dose) and Study Days 1, 2 and 3
  Laser Doppler flowmetry measures changes in red cell flux using a probe that scans a fixed volume of tissue, an indirect measure of flow can be obtained. Participants were examined in the left lateral position with no prior bowel preparation. The laser Doppler probe (DRT4 laser Doppler flow meter) was then placed against the rectal mucosa 10 centimeter above the lower limit of the anal margin, and pre-stress readings were taken after a period of 10 minutes of acclimatization in a room with an ambient temperature of 22 degrees Celsius. The dichotomous listening test was used as a psychological stressor. At the onset of stress, folk music was played into one ear and rock music into the other ear for 10 minutes. Readings were then taken during pre-stress and at 5-minute intervals during the stress and recovery periods. Baseline was defined as the pre-dose assessment. Change from Baseline was calculated by subtracting the Baseline value minus the post-randomization value.

SECONDARY OUTCOMES:
Number of participants with adverse events (AE) and serious adverse events (SAE) | Up to Week 14
  An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, may jeopardize the participant or require medical or surgical intervention to prevent one of the other outcomes listed in the definition above, or is an event of possible drug-induced liver injury.
Number of participants with abnormal clinical chemistry data of clinical concern | Up to Week 14
  The clinical chemistry parameters included albumin, calcium low, creatinine, glucose, magnesium, phosphorus, potassium, sodium, and bicarbonate. The total number of participants with clinical chemistry data of clinical concern have been presented.
Number of participants with abnormal hematology data of clinical concern | Up to Week 14
  The hematology parameters included white blood cell count, neutrophil count, hemoglobin, hematocrit, platelet count and lymphocytes. The total number of participants with hematology of clinical concern have been presented.
Participant perceived stress as assessed by a Visual Analogue Scale | Study Days 1, 2 and 3
  The acute emotional response to stress during each study visit was assessed using a 10 cm description-anchored visual analogue scale, ranging from 0 to 10, where 0=no-stress and 10=Most stressed ever. Higher scores indicated significant stress. Participants were asked to mark this before onset of stress, after 10 minutes of stress and finally after 10 minutes of recovery. After the pre-stress recordings, the period of either physiological or psychological stress were commenced and continued for 10 minutes, followed by a period of recovery for a further 10 minutes.
Systemic autonomic nervous system response as assessed by systolic blood pressure (SBP) and diastolic blood pressure (SBP) | Up to Week 14
  As an indicator of change in systemic autonomic activity, blood pressure was measured pre-stress, after 10 minutes of stress and after 10 minutes of recovery using a Dinamap.
Systemic autonomic nervous system response as assessed by heart rate (HR). | Up to Week 14
  As an indicator of change in systemic autonomic activity, HR was measured pre-stress, after 10 minutes of stress and after 10 minutes of recovery using a Dinamap.
Percent change from Baseline in participant reported threshold for pain as a measure to assess Visceral (rectal) electro sensitivity | Baseline (pre-dose) and Study Days 1, 2 and 3
  Visceral (rectal) sensitivity to pain was measured using previously validated techniques. In brief, a 1-cm bipolar electrode (21L10) mounted on a 14-gauge Foley catheter was placed initially into the anal canal before the period of acclimatization. The stimulation parameters were set at 0.5-millisecond pulse width and 10-Hertz frequency for rectal measurements. The current was then increased slowly and the participants were asked to report when they felt it was painful (pain). Rectal measurements were made 8 cm above the anal verge. Measurements were made pre-stress, after 10 minutes of stress, and then after 10 minutes of recovery. The catheter remained in situ throughout the study but was moved from anal to rectal sites for the 2 measurements. Baseline was defined as the pre-dose assessment. Change from Baseline was calculated by subtracting the Baseline value minus the post-randomization value.
Percent change from Baseline in participant reported threshold for perception of an electrical stimulus as a measure to assess Visceral (rectal) electro sensitivity | Study Days 1, 2 and 3
  Visceral (rectal) sensitivity to perception was measured using previously validated techniques. In brief, a 1-cm bipolar electrode (21L10) mounted on a 14-gauge Foley catheter was placed initially into the anal canal before the period of acclimatization. The stimulation parameters were set at 0.5-millisecond pulse width and 10-Hertz frequency for rectal measurements. The current was then increased slowly and the participants will be asked to report when they were first aware of this (perception). Rectal measurements were made 8 centimeter above the anal verge. Measurements were made pre-stress, after 10 minutes of stress, and then after 10 minutes of recovery. The catheter remained in situ throughout the study but will be moved from anal to rectal sites for the 2 measurements. Baseline was defined as the pre-dose assessment. Change from Baseline was calculated by subtracting the Baseline value minus the post-randomization value.
Change from Baseline in RMBF at 90 minutes post-dose | Baseline (pre-dose) and Study Days 1, 2 and 3
  RMBF was measured in response to both physiologic and psychological stress. Pre-stress readings were taken after 10 minutes of acclimatization. Readings were taken during pre-stress collections and at 5 minutes intervals during the stress and recovery period.Baseline was defined as the pre-dose assessment. Change from Baseline was calculated by subtracting the Baseline value minus the post-randomization value.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom